CLINICAL TRIAL: NCT06446700
Title: Correlation Between Neck Pain and Visual Disturbances in Smartphone Users
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Saeed Atallah, Principal investigator, Cairo University
Other Study IDs: neck pain and vision
Record Dates: First submitted 2024-05-23; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Neck Pain; Visual Disturbances
Keywords: neck pain; vision; smartphone
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: neck disability index and visual functional questionnaire — participants complete the 2 questionnaire by an online form and paper
  Other Names: visual functional questionnaire

SUMMARY:
the goal of this study is to Investigate the correlation between neck pain and visual disturbances in smartphone users.

DETAILED DESCRIPTION:
Study design:

Cross-sectional observational analytical study design conducted on smartphone users 2- Subject selection 141 subjects (who are smartphone users) according to sample size calculation will be selected randomly to complete the neck disability index and visual functional questionnaire 25 version 2000

ELIGIBILITY:
Inclusion Criteria:

* 141 subjects who are smartphone users
* Age between 18 to 50 years
* Both genders are included
* Subjects Who put in more than 4 hours a day using smartphone
* Participants without systemic illnesses or physical deformities were also included
* Consent: Participants who provide informed consent to participate in the study.
* Neck disability index will be used to assess how your neck pain has affected your ability to manage in everyday life.
* Visual Functioning Questionnaire version 2000 will be used to assess vision-related quality of life

Exclusion Criteria:

* People with head and neck injuries
* eye diseases
* People with diabetic retinopathy
* who had refractive correction surgery
* psychiatric problems (depression)
* people with systemic illnesses or physical deformities
* people who have vision impairments and disabilities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: participants from universities and local population
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Neck disability index | 1 month
  Patient-completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation.
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.
  The NDI can be scored as a raw score or doubled and expressed as a percent. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'.
  Points summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage.
  0 points or 0% means: no activity limitations, 50 points or 100% means complete activity limitation. A higher score indicates more patient-rated disability.
Visual functional questionnare | 1 month
  The VFQ-25 consists of a base set of 25 vision targeted questions representing 11 vision-related constructs, plus an additional single-item general health rating question The VFQ-25 takes approximately 10 minutes on average to administer in the interviewer format. There is also a self-administered version of theSurvey.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Elgendy, Study Director — Professor
Locations (1):
- Yasmin Saeed Atallah, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No